CLINICAL TRIAL: NCT01398566
Title: Clinical Trial of a Novel Rehabilitation Game (Phase I - Feasibility)
Brief Title: Clinical Trial of a Rehabilitation Game - SuperBetter
Acronym: SuperBetter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Lise Worthen-Chaudhari, Research Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011H0077
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Concussion; Mild Traumatic Brain Injury; Moderate Traumatic Brain Injury
Keywords: TBI; concussion; brain injury
MeSH Terms: conditions — Brain Concussion; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SuperBetter Play (Experimental): members of this group will play SuperBetter for 6 weeks (averaging 10 min per day of play for 6 week period)
  Interventions: Behavioral: SuperBetter play

INTERVENTIONS:
Behavioral: SuperBetter play — average 10 min of game play per day for 6 week period

SUMMARY:
Today's hospitals need innovative solutions to help patients transition from our care to self-management at home. The vast majority of the patients seen in Dodd Rehabilitation Hospital and associated clinics leave our care with persistent and life-altering challenges - behavioral, cognitive, emotional and/or physical. The period of time immediately following discharge is an under-addressed stage within the continuum of care. The investigators are researching solutions to help patients in this transition to self-care and believe that multiplayer gaming paradigms may be a promising innovation to facilitate this transition.

The investigators believe that Dr. Jane McGonigal's SuperBetter, and positive play games like it, are promising novel interventions that could make a positive difference in the ability of our patients to successfully transition to self care after discharge from therapeutic care.

Specifically, the investigators will evaluate feasibility of use of such a game by mild to moderate brain injured individuals and to record pilot data to help us plan a clinical effectiveness follow up study. Our goal is to finish this study with an intervention tailored for use within the clinical continuum of care and sufficient pilot data to prepare for a randomized clinical control trial of this intervention.

DETAILED DESCRIPTION:
Today's hospitals need innovative solutions to help patients transition from our care to self-management at home. The vast majority of the patients seen in Dodd Rehabilitation Hospital and associated clinics leave our care with persistent and life-altering challenges - behavioral, cognitive, emotional and/or physical. The period of time immediately following discharge is an under-addressed stage within the continuum of care. The investigators are researching solutions to help patients in this transition to self-care and believe that multiplayer gaming paradigms may be a promising innovation to facilitate this transition for several reasons:

1. Games can bring the power of social networks and alternate reality to bear on the real world work of post-injury self-management.
2. Games can use a digital platform, enabling quantification of performance in ways that could provide clinically-relevant documentation for post-discharge follow up efforts including tele-rehabilitation.
3. Today's youth are gamers. The investigators aim to tailor our rehabilitative approaches to leverage the existing ability of our youth in this paradigm. In addition, Dr. Jane McGonigal reports in her book, Reality is Broken, that within another decade the majority of the world's population will likely be gamers. The investigators aim to anticipate this shift and be ready for it.
4. Affordable games have the potential to be cost-effective aids and improvements over standard medical care protocols.

Despite the promise of games to facilitate transitions from hospital care to self care, no clinical studies have been done to establish best practices for applying gaming for rehabilitative purposes within the specific window of time in which discharge from standard care happens. While some commercially available games exist for those interested in health self-improvement, through companies such as That Game Company, Nintendo, Xbox, only the Nintendo Wii system has undergone clinical testing to demonstrate feasibility of use within the hospital-based model of patient care. Without more such evidence, the investigators are unable to confidently offer such novel interventions for our patients.

A new game, SuperBetter (SuperBetter, LLC, Sausilito, CA), has been developed to employ both social networking and alternate reality theory to achieve rehabilitative goals. SuperBetter is most similar to Facebook or Twitter in that users, or "gamers", create an account, invite others to be within their network, and post short status update messages. There are two major differences between SuperBetter and Twitter or Facebook, however. One difference is that this rehabilitation game will not offer a public option. The only people who can see a user's posts and status updates will have been specifically invited by that gamer; people outside the invited network will have no ability to "friend" a gamer, meaning there is no way to request to become part of a user's network - you must be invited by the account holder. The second difference is that SuperBetter assigns points to a gamer for attaining health goals such as: remembering to take medications each day; avoiding circumstances that exacerbate symptoms; checking in with someone within your trusted network (i.e. reaching out to your loved ones for support). Points are also assigned for "epic wins" which are defined by the patient and amount to things he or she cannot do today but want to be able to do tomorrow; this includes short term wins like hanging out with friends/loved ones or long term wins like getting back to playing sports.

The investigators believe that McGonigal's SuperBetter, and positive play games like it, are promising novel interventions that could make a positive difference in the ability of our patients to successfully transition to self care after discharge from therapeutic care. The investigators are conducting Phase I clinical testing (feasibility) to determine whether such a rehabilitation game is appropriate for use with: mild traumatic brain injured children and teens.

Specifically, the investigators will evaluate feasibility of use of such a game by mild traumatic brain injured individuals and to record pilot data to help us plan a clinical effectiveness follow up study. Our goal is to finish this study with an intervention tailored for use within the clinical continuum of care and sufficient pilot data to prepare for a randomized clinical control trial of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients: between 15 and 25 years old
* diagnosed within the last year with at least one traumatic brain injury (mild or moderate)
* subjective report of less than complete recovery from the injury
* easy access to computer with internet access
* compatible web browser (such as the latest version of Internet Explorer, Chrome, Firefox or other as determined by developers)
* has a support giver (18 or over) who is willing to participate in this study also

Exclusion Criteria:

● history of substance abuse as self reported by patient or reported by support giver

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lise Worthen-Chaudhari, MFA,MS,CCRC, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Physical Medicine and Rehabilitation Department, Columbus, Ohio, United States

REFERENCES:
- See also: Sponsor website — http://superbetter.com/
- See also: Game designer website — http://janemcgonigal.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinic patients (aged 13-18 years) with physician-diagnosed concussion and unresolved symptoms at 3 weeks to 12 months post injury between 13 August 2014 and 9 December 2014 were screened and recruited.
Pre-assignment Details: Follow-up ended on 7 January 2015. Participants were excluded for premorbid learning disabilities, concurrent illness/injury at pre-test and complicated or atypical symptom presentation per treating clinician (e.g. symptoms incongruent with cognitive load).
Groups:
- Gaming: Members of this group will play SuperBetter in addition to standard medical care for persistent concussion symptoms
Period: Overall Study
Arm/Group | Gaming
Started (Enroll up to 20 participants) | 20 (20 enrolled)
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Gaming: Members of this group will play SuperBetter in addition to receiving standard medical care for persistent concussion symptoms
Arm/Group | Gaming
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 20
Region of Enrollment [Number; unit: participants]
  United States | 20
Number of participants with Sports Concussion Assessment Tool-3 (SCAT-3)Symptoms Score > 1 [Count of Participants; unit: Participants] — The SCAT-3 is patient-reported outcome measure. Participants rate the severity level at which they are experiencing 22-items, that represent specific concussion symptoms. Severity per item ranges from 0 (none) to 6 (severe) at time of ecological momentary assessment. Scores are summed such that 0 corresponds to no symptoms, while 132 corresponds to severe incidence of all 22 items (i.e., worst presentation imaginable). Inclusion criteria for enrollment = a score of greater than 1.
  Participants | 20

OUTCOME MEASURES:

1. Primary Outcome: Participation
Description: Number of Participants who used the app and returned for post testing
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Gaming
Number analyzed (Participants) | 20
Participants | 14

2. Secondary Outcome: Satisfaction With App
Description: Satisfaction rating on a 7 point Likert scale ranging from 1 (very satisfied) to 7 (very dissatisfied) among those who used the app and returned for post testing
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Gaming
Number analyzed (Participants) | 14
units on a scale | 2.0 [2.0 to 2.0]

ADVERSE EVENTS:
Time Frame: 5 months (8/13/14 - 1/7/15)
Arm/Group | Gaming
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No